CLINICAL TRIAL: NCT01437007
Title: A Phase 1 Dose Escalation Study of Hepatic Intra-Arterial Administration of TKM 080301 (Lipid Nanoparticles Containing siRNA Against the PLK1 Gene Product) in Patients With Colorectal, Pancreas, Gastric, Breast, Ovarian and Esophageal Cancers With Hepatic
Brief Title: TKM 080301 for Primary or Secondary Liver Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110240; 11-C-0240
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2012-10-09

CONDITIONS: Colorectal Cancer With Hepatic Metastases; Pancreas Cancer With Hepatic Metastase; Gastric Cancer With Hepatic Metastase; Breast Cancer With Hepatic Metastase; Ovarian Cancer With Hepatic Metastase
Keywords: SNALP; Regional Therapy; Stage IV Disease; Adenocarcinoma; Unresectable; Liver Metastases; Colorectal Cancer; Stomach Cancer; Gastric Cancer; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Liver Cancer
MeSH Terms: conditions — Disease; Adenocarcinoma; Colorectal Neoplasms; Stomach Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Liver Neoplasms | interventions — TKM-080301

INTERVENTIONS:
Drug: TKM-080301

SUMMARY:
Background:

Cancer in the liver can start in the liver (e.g., primary liver cancer or hepatocellular cancer) or spread to the liver from cancers in other parts of the body (e.g. colon, pancreas, gastric, breast, ovarian, esophageal cancers, cancer with metastases to the liver.) People who have tumors that can be removed by surgery live longer than those whose cancer cannot be removed. Chemotherapy can shrink some tumors in the liver, which also helps people to live longer, and sometimes chemotherapy can shrink tumors enough that they can be removed by surgery. However, most chemotherapy drugs do not work well on tumors in the liver. In this study we are testing a new drug, TKM-080301, given directly into the cancer blood supply in the liver circulation, to see if it will cause tumors to shrink.

Objectives:

- To test the safety and effectiveness of TKM-080301 for cancer in the liver that has not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have inoperable cancer that has started in or spread to the liver.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood tests, and imaging studies.
* Participants will have a liver angiogram (type of X-ray study) to look at the blood flow in the liver and to place a catheter for delivery of the TKM080301.
* Participants will have a single dose of TKM-080301 given directly into the liver. After the drug has been given, the catheter will be removed. They will have frequent blood tests and keep a diary to record side effects.
* Participants may have two more doses, each dose given 2 weeks apart. {Before each dose, participants will have another angiogram and catheter placement.}They may also have liver biopsies to study the tumors.
* Two weeks after the third treatment (one full course), participants will have a physical exam, blood tests, and imaging studies. If the tumor is shrinking, they may have up to three more courses of the study drug.
* Participants will have follow up visits every 3 months for 2 years after the last course and then every 6 months as required.

DETAILED DESCRIPTION:
BACKGROUND:

- Metastatic liver disease is a life-limiting factor for patients with a variety of cancers. For

unresectable liver metastases, the 5-year survival is < 5%.

* For selected histologies the 5-year survival of resectable hepatic metastases ranges from 20-60%, suggesting that control of liver metastases could result in prolonged survival.
* Phase I through III trials have shown that Hepatic Arterial Infusion (HAI) is safe. However, agents used thus far in HAI have limited efficacy.
* TKM-080301 is a lipid nanoparticle (LNP) formulation containing siRNA against the PLK1 (polo-like kinase-1) gene product. More specifically, TKM-080301 is a type of LNP formulation, referred to as SNALP (Stable Nucleic Acid Lipid Particles). PLK1 has been validated as a molecular target and a prognostic factor in a variety of cancers. Inhibition of PLK1 activity in proliferating cancer cells rapidly induces mitotic arrest and apoptosis.
* This study will offer HAI with TKM-080301 to patients with unresectable and/or life threatening primary liver cancer or liver metastases.

OBJECTIVES:

Primary Objective:

- To evaluate feasibility of administering TKM-080301 via HAI and to characterize the pharmacokinetics (PK) and pharmacodynamics of TKM-080301 administered by HAI.

Secondary Objectives:

* To establish the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of TKM-080301.
* To evaluate response rate using RECIST, PET and EASL criteria.
* To evaluate the conversion rate from unresectable to resectable disease.

ELIGIBILITY:

* Patients with unresectable colorectal, pancreas, gastric, breast, ovarian and esophageal cancers with hepatic metastases; or primary liver cancer patients who have demonstrated progressive disease following standard of care treatment.
* 18 years old or greater with an ECOG 0-2
* Laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to surgery or chemotherapy.

DESIGN:

- This is a dose escalation phase-I study testing HAI of TKM-080301 for patients with

unresectable colorectal, pancreas, gastric, breast, ovarian and esophageal cancers with hepatic metastases, or primary liver cancers.

* Up to 54 patients who meet eligibility criteria will receive HAI with TKM-080301.
* Initial dose will be 4 mg/m(2); treatment will be given every 2 weeks for up to 12 doses.
* Patients will be evaluated every 6 weeks. Patients whose tumors become resectable will be offered this option; patients who show progressive disease will be taken off treatment. All patients will be followed for survival.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Histologically or cytologically confirmed colorectal, pancreas, gastric, breast, ovarian and esophageal cancers with hepatic metastases, or primary liver cancers (Hepatocellular carcinoma and Cholangiocarcinoma).
2. Hepatic disease must be measurable per RECIST Criteria (version 1.1).
3. Hepatic disease should be deemed unresectable as per standard of care criteria.

   Note: Evidence of limited unresectable extrahepatic disease on preoperative radiological studies is acceptable if the life-limiting component of progressive disease is in the liver.
4. All patients must have failed to respond to standard regimens or therapies known to provide clinical benefit. For example:

   - Patients with metastatic colorectal cancer must have received 5-FU and

   leucovorin in combination with either oxaliplatin and/or irinotecan, since level

   1 evidence support increase survival with these regimens, compared to 5-FU and leucovorin alone.

   - Patients with hepatocellular carcinoma must have received sorafenib, since level 1 evidence support increase survival.
5. Greater than or equal to 18 years of age
6. Must be able to understand and sign the Informed Consent Document
7. Clinical performance status of ECOG less than or equal to 2
8. Life expectancy of greater/equal than two months
9. Patients of both genders must be willing to practice birth control during and for four months after receiving chemotherapy
10. Hematology:

    * Absolute neutrophil count greater than or equal to 1500/mm(3) without the support of filgrastim.
    * Platelet count greater than or equal to 100,000/mm(3).
    * Hemoglobin greater than or equal to 9.0 g/dl.
11. Chemistry:

    * Serum ALT/AST less than or equal to 2.5 times the upper limit of normal.
    * Serum Albumin greater than or equal to 3.0 g/dL
    * Serum creatinine less than or equal to 1.5 times ULN unless the measured

    creatinine clearance is greater than 60 mL/min/1.73 m(2)

    - Total bilirubin less than or equal to 1.2 mg/dl
12. International Normalized Ratio (INR) less than or equal to 1.5
13. Seronegative for HIV antibody
14. No chemotherapy or any other investigational drugs within 4 weeks of treatment
15. LVEF greater than or equal to 50 percent
16. QT/QTc interval less than 450 ms

EXCLUSION CRITERIA:

1. Any known brain metastases (prior or current regardless of treatment status)
2. Women of child-bearing potential who are pregnant or breastfeeding, because of the potentially dangerous effects of the chemotherapy on the fetus or infant.
3. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune systems, recent myocardial infarction or heart failure (within 6 months of enrollment).
4. NYHA greater than or equal to 2
5. Childs B or C cirrhosis or with evidence of severe portal hypertension by history, endoscopy, or radiologic studies
6. Weight less than 40 kg
7. Significant ascites, greater than 1000cc in the absence of peritoneal disease
8. Concomitant medical problems that would place the patient at an unacceptable risk for the procedure/drug
9. Patient has known hypersensitivity or previous severe reactions to oligonucleotideor lipid-based products, including liposomal drug products (e.g. Doxil) and phospholipid-based products (parenteral nutrition, Intralipid)
10. Discretion of the PI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-08-26; Primary Completion 2012-06-21 (Actual); Study Completion 2012-06-21 (Actual)

PRIMARY OUTCOMES:
To evaluate feasibility of administering TKM-080301 via HAI, and establish MTD and DLT. | 2 years

SECONDARY OUTCOMES:
Characterize PK & pharmacodynamics of TKM 080301 | 2 years
Eval biological effects of TKM-080301 on biopsies performed before & after 1 cycle of tx | 2 years
To evaluate the potential conversion rate from unresectable to resectable disease. | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Steegmaier M, Hoffmann M, Baum A, Lenart P, Petronczki M, Krssak M, Gurtler U, Garin-Chesa P, Lieb S, Quant J, Grauert M, Adolf GR, Kraut N, Peters JM, Rettig WJ. BI 2536, a potent and selective inhibitor of polo-like kinase 1, inhibits tumor growth in vivo. Curr Biol. 2007 Feb 20;17(4):316-22. doi: 10.1016/j.cub.2006.12.037. Epub 2007 Feb 8. PMID 17291758
- [Background] Barr FA, Sillje HH, Nigg EA. Polo-like kinases and the orchestration of cell division. Nat Rev Mol Cell Biol. 2004 Jun;5(6):429-40. doi: 10.1038/nrm1401. No abstract available. PMID 15173822
- [Background] Strebhardt K, Ullrich A. Targeting polo-like kinase 1 for cancer therapy. Nat Rev Cancer. 2006 Apr;6(4):321-30. doi: 10.1038/nrc1841. PMID 16557283